CLINICAL TRIAL: NCT01949714
Title: Effect of Chronic Catecholamine Overproduction on Brown Adipose Tissue
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Esben Søndergaard, MD, PhD, Post Doc, University of Aarhus
Other Study IDs: ES-0005
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Pheochromocytoma; Adrenal Incidentaloma
MeSH Terms: conditions — Pheochromocytoma; Adrenal incidentaloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and adipose tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pheochromocytoma patients: Pheochromocytoma patients
  Interventions: Procedure: Removal of adrenal tumor

INTERVENTIONS:
Procedure: Removal of adrenal tumor

SUMMARY:
* To investigate the effect of catecholamine excess on brown fat.
* To evaluate the effect of brown fat on energy expenditure and lipid and glucose metabolism

ELIGIBILITY:
Inclusion Criteria:

* 10 patients with pheochromocytoma
* 5 patients with incidentaloma without hormone production
* Age > 18 years

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adrenal tumors
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
[18F]FDG uptake in brown adipose tissue | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology MEA, Aarhus Hospital, Aarhus C, Please Select, Denmark